CLINICAL TRIAL: NCT06095206
Title: to Evaluate the Pharmacokinetic Characteristics and Bioavailability of Recombinant Human Follicle Stimulating Hormone-CTP Fusion Protein Injection（GenSci094） in Healthy Male Subjects Before and After a Change in Manufacturing Site
Brief Title: The Pharmacokinetic and Bioavailability of GenSci094 Before and After a Change in Manufacturing Site
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Afﬁliated Hospital of North Sichuan Medical College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GenSci094-101
Record Dates: First submitted 2023-10-11; First posted 2023-10-23 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-12

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GenSci094 (Experimental): Participants received a single subcutaneous (SC) injection of 150 µg GenSci094 on day 1 pre-meal，PK and immunogenicity blood collection to day18， safety call follow-up completed at day 25
  Interventions: Drug: GenSci094

INTERVENTIONS:
Drug: GenSci094 — On the morning of day 1 pre-meal, a single SC injection of 150 μg GenSci094 was administered in the abdominal wall.

SUMMARY:
The bioavailability study is intended to evaluate the pharmacokinetic (PK) characteristics and the bioavailability of the two formulations in humans before and after the change of production site, in order to assess the possible impact of the site change on the pharmacokinetic characteristics of the drug and to clarify whether the two formulations are comparable before and after the change.

DETAILED DESCRIPTION:
This study used a single-center, open, randomized, single-dose, parallel-controlled trial design, and the study drug consisted of 1) the test drug (GenSci094 after the change in manufacturing site) and 2) the control drug (GenSci094 before the change in manufacturing site). Screened 48 healthy male subjects were randomly assigned to Group A (test drug) or Group B (control drug), randomized at timeprevious day（ D-1）, admitted to the Phase I clinical trial ward and put on a uniform diet; received 150 μg subcutaneous injection administration of the study drug on the following day (D1), and blood was collected for PK and immunogenicity up today 18（ D18）; and completed a safety telephone follow-up on day 25（D25）.

ELIGIBILITY:
Inclusion criteria

1. Subjects volunteered and signed an informed consent form and were able to understand and follow the trial requirements;
2. Healthy males aged 18-45 years old (including cut-off values);
3. Body weight ≥60kg and BMI between 19-28 kg/m2 (including cut-off values);
4. The subject's clinical history, physical examination, 12-lead electrocardiogram and laboratory tests during the screening period were not abnormal or the abnormalities were not clinically significant.
5. The subject agrees to use reliable contraception for himself/herself and his/her partner for the duration of the study and for a period of 3 months after study drug infusion.

Exclusion criteria

1. Persons with clinically significant metabolic/endocrine, hepatic, renal, hematologic, pulmonary, immunologic, cardiovascular, gastrointestinal, genitourinary, neurologic, or psychiatric disorders of any clinical severity or any other condition capable of interfering with the results of the test (at the discretion of the investigator) within the 3 months prior to the Screening Period and during the Screening Period;
2. Abnormalities in basic sex hormone tests of clinical significance (at the discretion of the investigator)
3. Abnormal liver function: alanine aminotransferase (ALT) or alanine transaminase (AST) > 1.5 times the upper limit of normal, or total bilirubin > 1.3 times the upper limit of normal;
4. Thromboembolic disease or history;
5. Those with a clear history of neurologic or psychiatric disorders (including epilepsy, dementia, depression or bipolar disorder, schizophrenia, etc.);
6. Prior history of gastrointestinal surgery, renal surgery, cholecystectomy, and other surgical procedures that, in the judgment of the investigator, may affect drug absorption or excretion;
7. Known history of allergy, anaphylaxis or hypersensitivity to the test preparation and any of its components or related agents;
8. Previous intolerance to phlebotomy/indwelling needle blood collection or history of blood or needle sickness;
9. Hypertension: systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg;
10. Positive screening tests for Hepatitis B Surface Antigen, Hepatitis C Virus Antibody, Human Immunodeficiency Virus (HIV) Antibody, or Treponema pallidum Antibody;
11. Those who have smoked >5 cigarettes per day in the 3 months prior to screening, or who are unable to abstain from the use of any tobacco-based products during the trial period;
12. Persons with drug dependence or drug abuse within 1 year prior to dosing, or who have a positive combined urine multi-drug test at check-in;
13. Those who have donated blood or lost ≥ 400 mL of blood within 3 months prior to the first dose; those who have difficulty collecting blood intravenously; and those who plan to donate blood during the trial or within 1 month of the end of the study;
14. Regular use of any prescription drug, over-the-counter drug, biologic, proprietary medicine, herbal medicine, vitamin dietary supplement or maintenance product, or vaccine within 2 weeks prior to the first dose, except for oral or buried long-acting contraceptives;
15. Persons who have been treated with any investigational drug or medical device in a clinical trial within 3 months prior to the first dose;

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Referring to the Chinese Pharmacopoeia 2020 edition of four general rules 9011 "Guidelines for human bioavailability and bioequivalence testing of pharmaceutical preparations", since GenSci094 is an FSH class drug, To ensure the safety of healthy female subjects, healthy males were selected as the subjects of this study to avoid GnRH agonist introduction and to reduce the risk of subjects, while only one dose of the drug was administered in this study and sex hormone was tested before and after the administration of the drug in male subjects
Enrollment: 48 (Actual)
Dates: Start 2023-09-19 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
Cmax（Maximum Serum Concentration of GenSci094(Cmax) | Venous blood was collected at 16 time points: 2h before, 6h, 12h, 24h, 30h, 36h, 48h (D3), 54h, 60h, 72h (D4), 96h (D5), 120h (D6), 192h (D9), 264h (D12), 336h (D15), and 408h (D18) for the determination of the concentration of GenSci094 in serum.
AUC0-t（（area under the time curve of blood concentration at time from 0 to the last time point selected | Venous blood was collected at 16 time points: 2h before, 6h, 12h, 24h, 30h, 36h, 48h (D3), 54h, 60h, 72h (D4), 96h (D5), 120h (D6), 192h (D9), 264h (D12), 336h (D15), and 408h (D18) for the determination of the concentration of GenSci094 in serum.]
AUC0-∞（Area Under the Serum Concentration-time Curve Extrapolated to Infinity [AUC(0-∞) | Venous blood was collected at 16 time points: 2h before, 6h, 12h, 24h, 30h, 36h, 48h (D3), 54h, 60h, 72h (D4), 96h (D5), 120h (D6), 192h (D9), 264h (D12), 336h (D15), and 408h (D18) for the determination of the concentration of GenSci094 in serum.
Tmax（Time to Reach a Maximum GenSci094 Serum Concentration (Tmax) | Venous blood was collected at 16 time points: 2h before, 6h, 12h, 24h, 30h, 36h, 48h (D3), 54h, 60h, 72h (D4), 96h (D5), 120h (D6), 192h (D9), 264h (D12), 336h (D15), and 408h (D18) for the determination of the concentration of GenSci094 in serum.
T1/2（GenSci094 Apparent Terminal Half-life (T1/2) | Venous blood was collected at 16 time points: 2h before, 6h, 12h, 24h, 30h, 36h, 48h (D3), 54h, 60h, 72h (D4), 96h (D5), 120h (D6), 192h (D9), 264h (D12), 336h (D15), and 408h (D18) for the determination of the concentration of GenSci094 in serum.
Safety and tolerability: Evaluation of safety through the adverse affects investigation | The entire study period begins when the subject signs the written ICF and ends with the completion of the last visit
Laboratory tests，physical examination，Post-medication results were analyzed for descriptive statistics on change from baseline values | 0-408hours
12-lead ECG：Heart rate, PR interval, QRS, QTc interval，Post-medication results were analyzed for descriptive statistics on change from baseline values | 0-408hours

SECONDARY OUTCOMES:
Immunogenicity: Anti-drug antibody (ADA) | Immunogenicity blood sample collection time points: within 1h before drug administration, 192h (D9), 408h (D18) for a total of 3 time points, and venous blood collected for serum immunogenicity analysis evaluation during early withdrawal visits]

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolan Yong, bachelor, Study Chair — chengdu xinhua hospital
Locations (1):
- Chengdu Xinhua Hospital, affiliated with Sichuan North Medical College, Chengdu, Sichuan, China